CLINICAL TRIAL: NCT06422624
Title: An Open Label, Single Dose, Dose Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of Semaglutide Extended-release Injectable Suspension in Normal Healthy, Adult, Human Study Participants Under Fasting Condition
Brief Title: A Study to Evaluate Safety, Tolerability and pK of Semaglutide ER Injectable Suspension in Healthy, Adult Human Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bostal Drug Delivery Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15403/23-24
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Semaglutide ER Injectable Suspension, 1 mg (Experimental): Participants receive a single of semaglutide ER injectable suspension at a lower dose 1 mg for safety, tolerability and pharmacokinetics assessements
  Interventions: Drug: Semaglutide Extended-release for Injectable Suspension, 1 mg
- Semaglutide ER Injectable Suspension, 4 mg (Experimental): Participants receive a single of semaglutide ER injectable suspension at a medium dose 4 mg for safety, tolerability and pharmacokinetics assessements
  Interventions: Drug: Semaglutide Extended-release for Injectable Suspension, 4 mg
- Semaglutide ER Injectable Suspension, 8 mg (Experimental): Participants receive a single of semaglutide ER injectable suspension at a higher dose 8 mg for safety, tolerability and pharmacokinetics assessements
  Interventions: Drug: Semaglutide Extended-release for Injectable Suspension, 8 mg

INTERVENTIONS:
Drug: Semaglutide Extended-release for Injectable Suspension, 1 mg — Singel-dose; Subcutaneous
  Arms: Semaglutide ER Injectable Suspension, 1 mg
Drug: Semaglutide Extended-release for Injectable Suspension, 4 mg — Singel-dose; Subcutaneous
  Arms: Semaglutide ER Injectable Suspension, 4 mg
Drug: Semaglutide Extended-release for Injectable Suspension, 8 mg — Singel-dose; Subcutaneous
  Arms: Semaglutide ER Injectable Suspension, 8 mg

SUMMARY:
The purpose of the trail is to evaluate the safety, tolerability and pharmacokinetics of a single escalated doses of semaglutide extended-release injectable suspension in healthy adult, human study participants under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

1. He/She should provide written informed consent.
2. He/She must be a healthy adult human male or non-pregnant, non-lactating females,18 - 45 years of age (both years inclusive).
3. He/She should have a body mass index ≥ 18.5 kg/m2 and ≤ 24.9 kg/m2 with body weight at least 55 kg for men and at least 48 kg for women.
4. He/She should have a baseline systolic blood pressure with upper limit of less than 140 mmHg and lower limit of more than or equal to 100 mm Hg. Similarly baseline diastolic blood pressure with upper limit less than 90 mm Hg and lower limit more than or equal to 60 mmHg.
5. He/She should have pulse rate not less than 60 beats/min and not more than 100 beats/min and respiratory rate not less than 14 breaths/min and not more than 18 breaths/min.
6. He/She must be of normal health as determined by medical history (including medication history) and physical examination performed within 21 days prior to the dosing.
7. He/She should have normal ECG, chest X-ray and vital signs.
8. He/She should have normal or clinically non-significant thyroid function tests (T3, T4 and TSH).
9. Availability of a study volunteer for the entire study duration and willingness to adhere to protocol requirements as evidenced by written informed consent.
10. If study volunteer is a female and is of child bearing potential practicing an acceptable method of birth control such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence for the duration of the study as judged by the investigator(s), or If she is postmenopausal with spontaneous amenorrhea for at least 01 year. or If she is surgically sterile (had a bilateral tubal ligation, bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 06 months).

Exclusion Criteria:

1. He/She is incapable of understanding the informed consent.
2. He/She has a history of hypersensitivity (e.g. anaphylactic reactions, angioedema and serious skin reactions) or idiosyncratic reaction to active or inactive ingredient in the Semaglutide extended-release injectable suspension or any other related drugs.
3. He/She has a history of impairment of renal, hepatic, cardiac, pulmonary or gastrointestinal function.
4. He/She has a history of tuberculosis, epilepsy, asthma, diabetes, psychosis and eye disorders.
5. He/She has history of any pulmonary disorder (COPD, Asthma, Bronchitis, other respiratory disorders) and skin related disorders.
6. He/She has a personal or family history of Medullary Thyroid Carcinoma (MTC) or any other thyroid tumors or Multiple Endocrine Neoplasia 2 (MEN 2) or any other endocrine disorders.
7. He/She has a history of pancreatitis, diabetic retinopathy, gall bladder disease.
8. He/She has undergone surgery within the past 3 months prior to screening, or those planning to undergo surgery during the trial period.
9. He/She has any difficulty in swallowing.
10. He/She regularly smokes more than 10 cigarettes daily or has difficulty in abstaining from tobacco for the entire study duration.
11. He/She has taken over the counter or prescribed medications, including vitamins, herbal supplements, insulin or drugs which promote insulin secretion, Sulfonylureas, any oral medications or any systemic medication within the past 30 days prior to dosing.
12. He/She has a history of any psychiatric illness, which may impair the ability to provide written, informed consent.
13. He/She has a history of alcohol or substance abuse within the last 05 years.
14. He/she using prohibited medications (e.g., sedative hypnotics, CNS depressants, including but not limited to opioid analgesics, benzodiazepines, sedating antidepressants or antipsychotics, sedating antiepileptic drugs, general anesthetics, muscle relaxants, and/or illicit CNS depressants).
15. He/She has clinically significant abnormal values of laboratory parameters.
16. He/She has participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 90 days.
17. He/She is unable to or unlikely to be compliant with protocol requirements or restrictions.
18. He/She, in whom study drug is contraindicated for medical reasons.
19. He/She is intolerant to venipuncture.
20. Positive results at screening for HIV, hepatitis B surface antigen (HBsAg), hepatitis C Virus (HCV) or syphilis.
21. Female volunteer who has used implanted or injected hormonal contraceptives anytime during the 06 months prior to study or used oral contraceptives within 14 days before dosing.
22. Female volunteer who demonstrates a positive pregnancy test.
23. Female study volunteer who is pregnant, breast-feeding or who is likely to become pregnant during the study.
24. Female using Hormonal IUD (Mirena), Norplant and other hormones, Depo-Provera, OCPs. (Females of child bearing age will be required to use 2 reliable forms of contraception such as condom and spermicidal or barrier method and spermicidal if sexually active. However, the use of Copper IUD or Tubal ligation are sufficient).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Cmax | From time zero up to the last time point with measurable concentration
  Maximum plasma concentration
AUC0-t | From time zero up to the last time point with measurable concentration
  Area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-inf | From time zero up to the last time point with measurable concentration
  Area under the plasma concentration-time curve from time zero to infinity